CLINICAL TRIAL: NCT03110120
Title: Interest of Serratus Plane Block in Postoperative Analgesia for Patients Undergoing Robot-assisted Mitral Valve Repair, MIDCAB or Partial Lung Resection
Brief Title: Interest of Serratus Plane Block in Postoperative Analgesia for Robot-assisted Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015/07JAN/008
Record Dates: First submitted 2017-03-08; First posted 2017-04-12 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-04

CONDITIONS: Analgesia; Robotic Surgery
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: Compare the efficacy of the serratus plane block with local infiltration after thoracic robot-assisted surgery
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient where randomized by the investigator after inform consent was signed The investigator prepared the syringes named "serratus" and "local" with levobupivacaine 0.25 or saline according to randomization The care provider injected the prepared syringes respectively in the serratus plane or locally without knowing their contents The outcome assessor evaluated the post operative pain and the 3 months followup without knowing the randomization
Oversight: Data Monitoring Committee: No

ARMS (2):
- serratus (Active Comparator): Serratus plane block and local control
  Interventions: Drug: 0.5% levobupivacaine injectable solution with 10 ml of physiological saline; Drug: 0.5% levobupivacaine injectable solution with physiological saline
- local (Sham Comparator): serratus control and local anesthesia
  Interventions: Drug: 0.5% levobupivacaine injectable solution with 10 ml of physiological saline; Drug: 0.5% levobupivacaine injectable solution with physiological saline

INTERVENTIONS:
Drug: 0.5% levobupivacaine injectable solution with 10 ml of physiological saline — Serratus plane block realized with a mixture of 10 ml of 0.5% levobupivacaine injectable solution with 10 ml of physiological saline
  Other Names: serratus plane block
  Arms: serratus
Drug: 0.5% levobupivacaine injectable solution with 10 ml of physiological saline — local infiltration of the wound with a mixture of 10 ml of 0.5% levobupivacaine injectable solution with 10 ml of physiological saline
  Other Names: local anesthesia
  Arms: local
Drug: 0.5% levobupivacaine injectable solution with physiological saline — Serratus plane block realized with 20 ml of injectable solution of physiological saline
  Other Names: local serratus
  Arms: local
Drug: 0.5% levobupivacaine injectable solution with physiological saline — local infiltration of the wound with 20 ml of injectable solution of physiological saline
  Other Names: local control
  Arms: serratus

SUMMARY:
The aim of the study is to compare the analgesia provided by the serratus plane block with local infiltration of the orifices of the trocars after thoracic robot-assisted surgery.

DETAILED DESCRIPTION:
In our hospital, the current practice to provide post operative analgesia for patients scheduled for robot-assisted mitral repair or oncological thoracic surgery is to dispense local anesthetics at the orifices of the trocars at the end of the surgery and to give a Patient Controlled Analgesia (PCA). Some of these patients are not comfortable and we observe a large percentage of chronic pain. Recently we tried to use the Serratus plane block realised before the beginning of the surgery, and it seemed that patients were more comfortable with a lower consumption of morphine. So we decided to perform a double blind, randomized study in this population of patients to compare the analgesia provided by the serratus plane block realized before the beginning of the surgery and the local infiltration of the wound at the end of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* mitral repair, coronary artery revascularization or thoracic surgery scheduled robot-assisted surgery

Exclusion Criteria:

* non robot-assisted surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
D0 pain intensity | 1 day
  Self reported pain intensity the day of surgery. Each item is scored 0-100 (0 - no pain, 100 - pain as bad as can be)

SECONDARY OUTCOMES:
D1 pain intensity | 3 days
  Self reported pain intensity the days after surgery. Each item is scored 0 - 100 (0 - no pain, 100 - pain as bad as can be)
morphine consumption | 5 days
  Consumption of morphine the day and 4 days after surgery as recorded on the PCA.
persistence of a chronic pain | 3 months
  Phone call 3 month after surgery to evaluate the persistence of pain

CONTACTS AND LOCATIONS:
Overall Officials: Christine Watremez, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Watremez Christine, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No